CLINICAL TRIAL: NCT04169542
Title: Potential Impact of the COVID -19 Pandemic on Financial Toxicity in Breast Cancer Surgical Patients: The Impact on Out of Pocket Costs, Lost Wages and Economic Strain
Brief Title: Impact of COVID-19 Pandemic on Out-of-Pocket Costs, Lost Wages, and Unemployment in Patients With Breast Cancer Undergoing Breast Surgery
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PA18-1077; NCI-2019-07463 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA18-1077 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Breast Ductal Carcinoma In Situ; COVID-19 Infection; Hereditary Breast Carcinoma; Invasive Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; COVID-19; Breast Cancer, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire): Patients complete up to 4 electronic questionnaires over 15 minutes before surgery and at 6, 12, and 24 months after surgery.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study investigates the impact of COVID-19 pandemic on out-of-pocket costs, lost wages, and unemployment in patients with breast cancer undergoing breast surgery. Post-mastectomy reconstructive patients are at high risk for financial toxicity (adverse effects of escalating health care cost on well-being). The goal of this study is to collect information about financial costs patients may have as a result of surgical treatment for cancer with or without breast reconstruction and to learn if COVID-19 affects patient costs of breast reconstruction. This may help researchers demonstrate the financial consequences of undergoing breast surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Obtain Comprehensive Score for financial Toxicity (COST) questionnaire data from the patients who are undergoing any form of mastectomy (with or without breast reconstruction).

II. To determine which patients are at higher risk of financial toxicity while pursuing breast reconstruction.

III. Assess if financial toxicity or distress is associated with worse BREAST-questionnaire (Q) performance as well as quality of life.

IV. Identify relationships between coronavirus disease 2019 (COVID-19) related productivity losses and financial toxicity.

OUTLINE:

Patients complete up to 4 electronic questionnaires over 15 minutes before surgery and at 6, 12, and 24 months after surgery.

After completion of study, patients will be followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Have an indication for surgical treatment of invasive breast cancer or ductal breast carcinoma in situ (DCIS) or prophylaxis in the setting of genetic mutations or strong family history
* English-speaking
* Able to complete consent
* Able to fill out computer survey material

Exclusion Criteria:

* Non-English-speaking
* Those with recurrent or metastatic disease or concurrent primary cancers
* Patients undergoing breast conservation therapy will also be excluded from the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are evaluated for breast reconstruction at MD Anderson Cancer Center (Texas Medical Center, Katy, League City, Memorial City, Sugar Land, The Woodlands) and, pending Institutional Review Board approval, domestic institutions in the MD Anderson Cancer Network
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-05-21 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of financial toxicity | Up to 1 year after completion of study
  Will be measured by the Comprehensive Score for financial Toxicity questionnaire. Summary statistics including mean, standard deviation, median, and range for continuous variables, and frequency count and percentage for categorical variables will be provided. Various subgroup analyses may occur. In these cases, continuous variables will be compared using the two-sample t-test and categorical variables will be compared using chi-squared test or Fisher's exact test. Multivariate regression analysis will be performed to account for confounding and to increase the robustness of any causal inference.

SECONDARY OUTCOMES:
Correlation between economic disruption from coronavirus disease 2019 (COVID-19) and financial toxicity | Up to 1 year after completion of study
  Summary statistics including mean, standard deviation, median, and range for continuous variables, and frequency count and percentage for categorical variables will be provided. Various subgroup analyses may occur. In these cases, continuous variables will be compared using the two sample t-test and categorical variables will be compared using chi-squared test or Fisher's exact test. Multivariate regression analysis will be performed to account for confounding and to increase the robustness of any causal inference.
Relationship between financial toxicity and patient reported quality of life | Up to 1 year after completion of study
  Will be assessed using the Short Form-12 survey. Summary statistics including mean, standard deviation, median, and range for continuous variables, and frequency count and percentage for categorical variables will be provided. Various subgroup analyses may occur. In these cases, continuous variables will be compared using the two-sample t-test and categorical variables will be compared using chi-squared test or Fisher's exact test. Multivariate regression analysis will be performed to account for confounding and to increase the robustness of any causal inference.
Relationship between financial toxicity and patient reported satisfaction with breast reconstruction | Up to 1 year after completion of study
  Will be assessed using the Breast-Q survey. Summary statistics including mean, standard deviation, median, and range for continuous variables, and frequency count and percentage for categorical variables will be provided. Various subgroup analyses may occur. In these cases, continuous variables will be compared using the two-sample t-test and categorical variables will be compared using chi-squared test or Fisher's exact test. Multivariate regression analysis will be performed to account for confounding and to increase the robustness of any causal inference.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Chu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas

REFERENCES:
- See also: http://www.mdanderson.org — http://www.mdanderson.org